CLINICAL TRIAL: NCT05040113
Title: A Clinical Study to Evaluate Absorption, Metabolism and Excretion of [14C] CBP-307 in Healthy Chinese Male Adult Subjects - Human Mass Balance and Biotransformation Study of [14C] CBP-307
Brief Title: A Study On Human Mass Balance And Biotransformation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Connect Biopharm LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CBP-307CN004
Record Dates: First submitted 2021-08-02; First posted 2021-09-10 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-01

CONDITIONS: Healthy Adult Subjects

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CBP-307 (Experimental): Take CBP-307orally at 30 min ± 2 min after the start of high-fat breakfast intake
  Interventions: Drug: CBP-307

INTERVENTIONS:
Drug: CBP-307 — CBP-307 capsules oral administration

SUMMARY:
This study will evaluate the absorption,metabolism and excretion of CBP-307 in healthy chinese male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. A healthy male adult
2. Age: 18 to 45 years old (inclusive)
3. Weight: body mass index (BMI) is between 19 and 26 kg/m2(inclusive), and weight of no less than 50 kg
4. Subjects who are willing to sign Informed Consent Form
5. Subjects should be able to communicate well with the investigator and be able to complete the study in accordance with the protocol

Exclusion Criteria:

-

Examinations:

1. Any abnormal and clinically significant findings to physical examination, vital sign, routine laboratory tests (such as hematology, blood chemistry, blood coagulation function, urinalysis, fecal occult blood), thyroid function test, 12-lead ECG, chest CT, abdominal B-ultrasonography (liver, gallbladder, pancreas, spleen and kidney) and so on
2. Heart rate at screening period < 60 bpm, or 12-lead ECG QTcF ≥450 msec
3. Anyone has positive examination result of HBsAg/HBeAg, HCV antibody, HIV antibody and treponema pallidum antibody
4. Screening for novel coronavirus infection: clinically significant abnormity of C-reactive protein, or positive novel coronavirus nucleic acid

   Medication history:
5. Use of any drug that inhibits or induces the function of hepatic drug-metabolizing enzymes within 30 days prior to screening (see Appendix 1)
6. Use of any prescription drugs, over-the-counter drugs, Chinese herbal medicines or food supplement such as vitamins, calcium supplement within 14 days prior to Screening
7. Use of any investigational drug within 3 months, or the drug withdrawal is less than 6 half-lives (whichever is longer) prior to successful enrollment for dosing

   Medical history and surgery history:
8. Any history of clinically serious disease, or presence of illness/condition that the investigator considers would affect the study results, including but not limited to the diseases of circulatory system, respiratory system, endocrine system, nervous system, digestive system, urinary system or history of blood, immune, mental and metabolic diseases
9. History of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmia, torsade ventricular tachycardia, ventricular tachycardia, AV block, QT prolongation syndrome, or QT prolongation symptoms and family history, indicated by genetic evidence or sudden death of a close relative due to cardiac conditions at a young age
10. Major surgery history or surgical incision does not completely heal within 6 months prior to the screening; Major surgery includes, but is not limited to, any subject with significant bleeding risk, prolonged general anesthesia, incision of a biopsy or significant traumatic injury
11. Allergic constitution, such as a known history of allergies to two or more substances; or may be allergic to the investigational product or its excipients based on the investigator's judgment
12. Suffering haemorrhoids or perianal disease with blood in the stool or regularly, irritable bowel syndrome, inflammatory bowel disease

    Life style:
13. Subjects have habitual constipation or diarrhoea
14. Subjects are alcoholism, or frequent alcohol consumption within six months prior to screening, which means drinking more than 14 units of alcohol every week (one unit alcohol equals 360 mL of beer, 45 mL of 40% alcohol or 150 mL of wine); or the alcohol breath test result is ≥20 mg/dl in screening
15. Subjects have smoked more than 5 cigarettes per day in three months before screening, or habitual use of nicotine products, and who can not quit smoking during the study
16. Abusing drug, using soft drugs such as marijuana three months prior to screening, or using hard drugs such as cocaine, amphetamine, phencyclidine, etc. one year prior to screening; or urine test for drugs is positive at screening
17. Subjects have habitual drinking of grapefruit juice, excessive tea, coffee and/or caffeinated beverages, and who can not be abstained during the study

    Others:
18. Subjects who have to work in radioactive conditions in long time, participated in radio-labeled drug clinical study or had significant radioactive exposure within one year before the study, no less than 2 times of chest/abdominal CT, or no less than 3 times of different types of X-ray exam
19. Subjects with a history of fear of needles, hemophobia, difficulty in blood collection or inability to tolerate venipuncture blood collection;
20. Subjects who plan to have children or donate sperm during the study period and within 1 year after completion of the study, or those who disagree to take strict contraceptive measures during the study or within 1 year after completion of the study for themselves or their spouses (see Appendix 3 for details)
21. Subjects who received any vaccine within 4 weeks before screening, or plan to receive the vaccine during the study
22. Subjects, who have had blood loss/donation up to 400 mL within 3 months, or received blood transfusion within 1 month prior to screening
23. Subjects determined by the investigators to be unsuitable for participating in this study for any reasons

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-09-04 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | Pre-dose and 1hour,2hour,4hour,6hour,7hour,8hour,10hour,12hour,24hour,48hour,72hour,96hour,120hour,144hour,168hour,216hour,264hour,312hour,360hour,408hour,456hour,504hour post-dose
  Ratio of total radioactivity in whole blood to that in plasma
Cumulative recovery of total radioactivity in urine or/and feces | -24 to 0 hour predose to Day22
  Percentage of each metabolite in urine and feces to the administered dose (% of administered dose) or percentage of circulating metabolites in plasma to total exposure AUC (% AUC)
Time to Peak (Tmax) | Pre-dose and 1hour,2hour,4hour,6hour,7hour,8hour,10hour,12hour,24hour,48hour,72hour,96hour,120hour,144hour,168hour,216hour,264hour,312hour,360hour,408hour,456hour,504hour post-dose
  Ratio of total radioactivity in whole blood to that in plasma
Area under the curve (AUC0-t and AUC0-inf) | Pre-dose and 1hour,2hour,4hour,6hour,7hour,8hour,10hour,12hour,24hour,48hour,72hour,96hour,120hour,144hour,168hour,216hour,264hour,312hour,360hour,408hour,456hour,504hour post-dose
  Ratio of total radioactivity in whole blood to that in plasma
Elimination half-life (t1/2) | Pre-dose and 1hour,2hour,4hour,6hour,7hour,8hour,10hour,12hour,24hour,48hour,72hour,96hour,120hour,144hour,168hour,216hour,264hour,312hour,360hour,408hour,456hour,504hour post-dose
  Ratio of total radioactivity in whole blood to that in plasma
Apparent Clearance (CL/F) | Pre-dose and 1hour,2hour,4hour,6hour,7hour,8hour,10hour,12hour,24hour,48hour,72hour,96hour,120hour,144hour,168hour,216hour,264hour,312hour,360hour,408hour,456hour,504hour post-dose
  Ratio of total radioactivity in whole blood to that in plasma
Apparent Volume of Distribution (Vd/F) | Pre-dose and 1hour,2hour,4hour,6hour,7hour,8hour,10hour,12hour,24hour,48hour,72hour,96hour,120hour,144hour,168hour,216hour,264hour,312hour,360hour,408hour,456hour,504hour post-dose
  Ratio of total radioactivity in whole blood to that in plasma
Mean Residence Time (MRT) | Pre-dose and 1hour,2hour,4hour,6hour,7hour,8hour,10hour,12hour,24hour,48hour,72hour,96hour,120hour,144hour,168hour,216hour,264hour,312hour,360hour,408hour,456hour,504hour post-dose
  Ratio of total radioactivity in whole blood to that in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Suzhou Connect, Study Director — Connect Biopharm LLC
Locations (1):
- Connect Investigative Site, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No